CLINICAL TRIAL: NCT02684019
Title: Goal Directed Propofol Sedation With Magnesium Sulphate Versus Dexmedetomidine for ERCP Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, khalda G Moustafa, Professor of anesthesiology, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TBRI project (code number111A)
Record Dates: First submitted 2016-02-06; First posted 2016-02-17 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Lack of Drug Action
Keywords: Endoscopic retrograde cholangiopancreatography; sedation; dexmedetomidine; propofol; Magnesium sulphate; Bispectral index monitoring
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Group M: the Drug consisted of 2 ampoules each one containing 2500 mg magnesium sulphate (Egypt Otsuka pharma.Co)in 50 ml syringe .(i.e. 100 mg/ml). Loading dose was 40mg/kg, given over 10min and maintenance dose was 10mg/kg/h.
  Group D: the Drug consisted of 2ml containing 200μg Dexmedetomidine (precedex®; united pharmaceutical group company, USA) diluted up to 50ml with normal saline (4μg/ml). Loading dose was 1μg/kg; given over 10min. The maintenance dose was 0.5 μg / kg / h.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): 1microgram/kilogram loading dose followed by 0.5 microgram/kilogram/hour IV
  Interventions: Drug: Dexmedetomidine
- Magnesium sulphate (Active Comparator): 40milligram/kilogram loading dose followed by 10milligram/kilogram/hour IV
  Interventions: Drug: Magnesium Sulphate

INTERVENTIONS:
Drug: Dexmedetomidine — added to propofol sedation
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Magnesium Sulphate — added to propofol sedation
  Arms: Magnesium sulphate

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an invasive longer endoscopic procedure. It is performed in remote locations under a continuum of anesthetic depth, ranging from conscious to deep sedation leading to general anesthesia.

Propofol sedation for (ERCP) procedures is the most popular current technique that has generated controversy in the medical field. Propofol can be safely administered because of its shorter half-life which results in a shorter recovery time than conventional sedation (opioid and/or benzodiazepine) that makes it widely used for sedation in many gastrointestinal procedures including ERCP. However, because of its narrow therapeutic window, the level of conscious sedation can easily go deeper from moderately deep sedation to near general anesthesia. Therefore, propofol as a sole agent can cause oversedation and apnea. Depth of sedation could be estimated better when target effect concentration of propofol is titrated by using bispectral index monitoring device(BIS).Targeting BIS within a specific range ensures additional safety during the procedure. Scores between 60-80 have been recommended for sedation. Propofol requirement can be reduced with addition of adjuvants (eg. Ketamine, Magnesium sulfate and Dexmedetomidine). Most adjuncts have analgesic properties with opioid and anesthetic sparing effects, without clinically significant respiratory depression.

Dexmedetomidine, is a selective alpha 2 agonist; it has sedative, amnestic, and analgesic properties. It is a useful addition to a propofol/remifentanil anesthetic combination as it reduced their requirements intraoperatively and can help supplement analgesia postoperatively. Its combination with propofol was proved to provide satisfactory anesthesia for upper gastrointestinal (GI)) endoscopy in obstructive sleep apnea patients .

Magnesium can also act as an adjuvant in analgesia due to its properties as calcium channel blocker and N-methyl-D-aspartate antagonists .It was suggested to be a near ideal intravenous (IV) adjunct to propofol/ remifentanil based total anesthesia in gynaecology patients .

Hypothesis of this study is that Magnesium sulfate can have a propofol sparing effect during ERCP procedures guided by BIS monitoring as efficient as dexmedetomidine but with less cost and complications together with more patient and doctor satisfaction in addition to better patient outcome.

DETAILED DESCRIPTION:
After Theodor Bilharz Research Institute (TBRI) Ethics Committee approval, sixty patients scheduled for ERCP procedures will be informed about the study and written consents will be obtained.

Patients will be allocated into two groups, thirty patients each, Magnesium (M) and Dexmedetomidine (D). Group (M) will receive 40 mg.kg-1 of magnesium sulphate bolus followed by IV infusion of 10 mg.kg-1.h-1. Group (D) will receive dexmedetomidine bolus (1μg.kg-1) followed by infusion of 0.5μg.kg-1h-1 all through the procedure.

Randomization of the patients will be established by computer generated random number table utilizing sealed envelope technique.

On arrival to the ERCP suit, two IV cannulae will be inserted in both hands of each patient in both groups. One for isotonic saline infusion and propofol administration and the other will be preserved for the study drug administration. IV fluid will be started at a rate of 8-12 ml.kg-1.h-1 continued throughout the procedure. All patients will be premedicated with intravenous pantoprazole 40mg and ondansetron 8mg.

Routine monitoring of ECG, pulse oximetry, non-invasive blood pressure will be established before induction of sedation. BIS three electrodes sensor will be applied over the patient's forehead using fronto-temporal montage for the monitoring of level of sedation . The baseline variables will be recorded and documented as well as continuous monitoring and documentation every 5 min for the first 30 min and every 10 min till the end of procedure. Supplemental oxygen will be administered with nasal prongs at 3 l.min-1. The total duration of the procedure, defined as the time taken from insertion of the endoscope to its removal, will also be documented.

Each study drug will be loaded in 50 ml syringes (for both bolus and infusion) & labeled as "study drug bolus" and "study drug infusion". The identity of the constituted drug in the syringe is not revealed to the anesthetist handling the patients and the observer recording the post procedure variables. Depending upon the body weight, each patient will receive a bolus of the study drug, diluted up to 50 ml with saline (direct IV)followed by infusion of the same drug in another 50 ml using a syringe pump. Each bolus will be given and the rate of drug infusion will be adjusted by the anesthesia resident not involved in the study.

The study drugs IV infusions will be administered using injector pumps with unidentified screen to assure that the observer remains blinded.

For each patient, bolus dose of the each study drug will be administered slowly over 10 min, after mouth gag insertion and patient positioning (either lateral or prone position) followed by induction with propofol in a dose of 0.5-1.5 mgkg-1, targeting BIS between 60-70.Once the target BIS is attained, the infusion of the study drug is started with the pre-adjusted rate (discussed before) along with the propofol maintenance infusion starting at a rate of 3 mg/kg/hr to be adjusted to maintain a BIS value between 60-70.At the end of the procedure, propofol and study drug infusions will be stopped. BIS values will be allowed equilibrating above 80. Patients oropharynx will be thoroughly suctioned and patients will be turned supine with head up tilt (15 degrees), to allow for complete recovery with eye opening on command, ability to handle secretions, follow simple commands, hemodynamic stability, maintaining O2 saturation at room air >95% and attainment of BIS value >90 as end points

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I, II or III.
* Body mass index (BMI) ˂30
* Patients scheduled for ERCP procedures

Exclusion Criteria:

1. Obesity (BMI >30)
2. Evidence of hepatic encephalopathy, ascites.
3. Sever renal, endocrine and respiratory dysfunction.
4. Atrioventricular conductance disturbance.
5. Symptomatic bradycardia <35 bpm
6. Hemodynamically unstable patients on inotropic support.
7. Neurological disorders
8. Myasthenia gravis.
9. Hypo/Hyperkalemia (Potassium <3meq/l or>5.5meq/l) (risk of dysrhythmias).
10. Chronic treatment with calcium channel blockers or magnesium
11. Opioid or analgesic abuse
12. Allergy to Propofol/ egg or any other study drugs.
13. Pregnancy and lactation

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Total propofol consumption | through study completion, an average of one hour
  0.5-1.5 mg as induction dose guided by bispectral index between 60-70 followed by infusion ranged from 3-5 mg/kg/h keeping BIS between 60-70

SECONDARY OUTCOMES:
Mean arterial blood pressure | through study completion, an average of one hour
  Every 5 min for the first 30 min and every 10 min till the end of procedure.Every 15 min in post-anesthesia care unit
Time to discharge | 15 minutes
  Time to reach modified Aldrete score more than 9
Cost | through study completion , an average of one hour
  The sum of all the drugs costs
Complication and side effects | through study completion , an average of one hour
  dizziness, vomiting or headache
Heart rate | through study completion, an average of one hour
  Every 5 min for the first 30 min and every 10 min till the end of procedure.Every 15 min in post-anesthesia care unit

OTHER OUTCOMES:
Patient satisfaction | through study completion, an average of one hour
  10 point numeric scale
Doctor satisfaction | through study completion, an average of one hour
  10 point numeric scale

CONTACTS AND LOCATIONS:
Overall Officials: Hend H Kamel, Professor, Study Chair — Theodor Bilharz Research Institute; Maher F Mahmoud, Professor, Study Chair — Kasr El Aini hospital,Faculty of medicine, Cairo University,; Eslam A Mohamed, Lecturer, Principal Investigator — Kasr El Aini hospital,Faculty of medicine, Cairo University,; Nabaweya M Kamal, Professor, Study Director — Theodor Bilharz Research Institute; Mohammed A Maher, Lecturer, Principal Investigator — Theodor Bilharz Research Institute; Ahmed S Abd El Azeem, Residant, Principal Investigator — Theodor Bilharz Research Institute; Khalda G Radwan, Professor, Study Director — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jeurnink SM, Steyerberg E, Kuipers E, Siersema P. The burden of endoscopic retrograde cholangiopancreatography (ERCP) performed with the patient under conscious sedation. Surg Endosc. 2012 Aug;26(8):2213-9. doi: 10.1007/s00464-012-2162-2. PMID 22302536
- [Result] Ramkiran S, Iyer SS, Dharmavaram S, Mohan CV, Balekudru A, Kunnavil R. BIS Targeted Propofol Sparing Effects of Dexmedetomidine Versus Ketamine in Outpatient ERCP: A Prospective Randomised Controlled Trial. J Clin Diagn Res. 2015 May;9(5):UC07-12. doi: 10.7860/JCDR/2015/12435.5991. Epub 2015 May 1. PMID 26155536
- [Result] Fluhr G, Mayerle J, Weber E, Aghdassi A, Simon P, Gress T, Seufferlein T, Mossner J, Stallmach A, Rosch T, Muller M, Siegmund B, Buchner-Steudel P, Zuber-Jerger I, Kantowski M, Hoffmeister A, Rosendahl J, Linhart T, Maul J, Czako L, Hegyi P, Kraft M, Engel G, Kohlmann T, Glitsch A, Pickartz T, Budde C, Nitsche C, Storck K, Lerch MM. Pre-study protocol MagPEP: a multicentre randomized controlled trial of magnesium sulphate in the prevention of post-ERCP pancreatitis. BMC Gastroenterol. 2013 Jan 15;13:11. doi: 10.1186/1471-230X-13-11. PMID 23320650
- [Result] James MF. Clinical use of magnesium infusions in anesthesia. Anesth Analg. 1992 Jan;74(1):129-36. doi: 10.1213/00000539-199201000-00021. No abstract available. PMID 1734773
- [Result] Wang D, Chen C, Chen J, Xu Y, Wang L, Zhu Z, Deng D, Chen J, Long A, Tang D, Liu J. The use of propofol as a sedative agent in gastrointestinal endoscopy: a meta-analysis. PLoS One. 2013;8(1):e53311. doi: 10.1371/journal.pone.0053311. Epub 2013 Jan 8. PMID 23308191
- [Result] Mukhopadhyay S, Niyogi M, Sarkar J, Mukhopadhyay BS, Halder SK. The dexmedetomidine "augmented" sedato analgesic cocktail: An effective approach for sedation in prolonged endoscopic retrograde cholangio-pancreatography. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):201-6. doi: 10.4103/0970-9185.155149. PMID 25948901